CLINICAL TRIAL: NCT03000491
Title: Developing a National Learning Health System for Asthma to Reduce the Risk of Asthma Attacks and the Risk of Asthma Hospitalisations and Deaths
Brief Title: Learning Health System for Asthma
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC16078
Record Dates: First submitted 2016-09-06; First posted 2016-12-22 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2016-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — Variations in clinical practice as assessed by data relating to asthma extracted from patient electronic health records.
  Other Names: ID: AC16078 NCT03000491

SUMMARY:
This study forms an initial phase of work aimed at developing a learning health system (LHS), whereby data relating to asthma is extracted from patient electronic health records (EHRs) across Scotland, analysed to explore variations in clinical practice and then shared with general practices to highlight any improvements that can be made so that they can better support people with asthma.

If successful, the investigators hope to progress to the main quality improvement phase involving an increased number of practices and then incrementally build this up to cover the whole of Scotland.

DETAILED DESCRIPTION:
The UK has amongst the highest rates of asthma in the world as well as some of the poorest health outcomes from asthma.

Investigations into asthma deaths in the UK have found that the way patients were managed in the time leading up to their death could be improved significantly and half of asthma deaths are potentially avoidable. For most people with asthma, symptoms can come and go and sometimes be erratic. To prevent these symptoms, there is a window of opportunity to intervene with the appropriate care. This window occurs between when someone experiences early symptoms like night cough or wheeze and when they experience a full-blown asthma attack.

Most people with asthma receive care primarily in their general practice. General practices have a history of using health information technology to care for their patients. The use of this technology over time has resulted in the creation of rich electronic healthcare data. Through this rich data there are opportunities to create a system whereby clinical management can be benchmarked and improvements highlighted.

This study forms an initial phase of work aimed at developing a learning health system (LHS), whereby data relating to asthma is extracted from patient electronic health records (EHRs) across Scotland, analysed to explore variations in clinical practice and then shared with general practices to highlight any improvements that can be made so that they can better support people with asthma.

If successful, the investigators hope to progress to the main quality improvement phase involving an increased number of practices and then incrementally build this up to cover the whole of Scotland.

ELIGIBILITY:
Inclusion Criteria:

• Patients registered with general practices across Scotland.

Exclusion Criteria:

* Patients from general practices that do not to opt-in to the study.
* Patients with a READ code recording dissent from use of their records for research purposes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (with and without asthma) in Scotland registered with primary care practices from 2010-2015.
Sampling Method: Non-Probability Sample
Enrollment: 750000 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Variations in clinical practice as assessed by data relating to asthma extracted from patient electronic health records. | At study completion (3 months)
  Variations in clinical practice as assessed by data relating to asthma extracted from patient electronic health records.

CONTACTS AND LOCATIONS:
Locations (1):
- University ot Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No